CLINICAL TRIAL: NCT05257668
Title: The Effect of Intradialytic High-Intensity Interval Training and Moderate Intensity Training on Dialysis Adequacy and Functional Capacity in Hemodialysis Patients
Brief Title: Intradialytic High-Intensity Interval Training in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin ASLAN KELEŞ (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Yasemin ASLAN KELEŞ, Physiotherapist, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intradialytic HIIT
Record Dates: First submitted 2021-11-30; First posted 2022-02-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: End Stage Renal Disease; Exercise, Compulsive
Keywords: intradialytic exercise; high-intensity interval training; chronic kidney disease; dialysis adequacy; functional capacity
MeSH Terms: conditions — Kidney Failure, Chronic; Compulsive Exercise; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): High intensity interval training
  Interventions: Other: High Intensity Interval Exercise Training
- Group 2 (Active Comparator): Moderate intensity training
  Interventions: Other: Moderate Intensity Exercise Training
- Group 3 (No Intervention): Control

INTERVENTIONS:
Other: High Intensity Interval Exercise Training — High Intensity Interval Training Group
  Arms: Group 1
Other: Moderate Intensity Exercise Training — Moderate Intensity Training Group
  Arms: Group 2

SUMMARY:
Chronic Kidney Disease (CKD) is defined as a chronic, progressive degeneration state in the regulation of the fluid-electrolyte balance of the kidney and metabolic-endocrine functions as a result of the glomerular filtration rate (GFR) falling below 60 ml/min/1.73 m², regardless of the etiology of the kidney disease. End Stage Renal Failure (ESRD) is the last stage of CRF and is a life-threatening condition. Although the majority of ESRD patients survive on dialysis, their quality of life and functional capacity decrease due to uremic cardiomyopathy, cardiovascular diseases, anemia, diabetes mellitus, bone diseases, deconditioning, fatigue, weakness, inactivity and accompanying psychological problems.

Rehabilitation program including exercise in CKD patients; The program, which is performed under observation on non-dialysis days, can be applied in three ways: the (intradialytic) rehabilitation program performed during hemodialysis in the dialysis unit, and the home exercise program. Intradialytic exercise (IDE) is defined as exercise training performed during the hemodialysis session to increase the patient's strength and endurance and thus target various physiological and psychosocial parameters. Three types of exercises are generally recommended in the exercise program for dialysis patients. These are aerobic exercise, strengthening exercise, and combined aerobic and resistance exercise program. Aerobic exercise (both on dialysis and on non-dialysis days) is the most common type of exercise used in hemodialysis patients. It is stated that physical exercise improves the exercise capacity, muscle strength, functional capacity and quality of life of patients receiving dialysis treatment, provides blood pressure control, reduces the risk of diabetes development and cardiovascular disease, alleviates depression and anxiety symptoms, increases survival and dialysis efficiency.

When the literature is examined, no study has been found that examines how the application of high-intensity intermittent exercise training, which has very important advantages, in the intradialytic process has an effect. Therefore, the aim of our study is to compare the effects of intradialytic high-intensity intermittent exercise training and moderate-intensity exercise training on dialysis effectiveness, functional capacity and quality of life in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-65
* Having Stage 5 (ESRD) CRF according to GFR
* Literate
* Cooperative
* Dialysis treatment for at least three months

Exclusion Criteria:

* History of myocardial ischemia in the last 6 months
* Uncontrollable diabetes mellitus,
* Uncontrollable hypertension
* Heart failure
* Malignant disease
* Mental retardation
* Illiteracy
* Uncooperative
* Neurological or orthopedic disability

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Dialysis Adequacy | 8 weeks
  Kt/V
6 Minute Walking Test | 8 weeks
  Functional Capacity
5X Sit-to-Stand Test | 8 weeks
  Functional Capacity
Kidney Disease Quality of Life-36 | 8 weeks
  Life Quality

SECONDARY OUTCOMES:
Beck Depression Scale | 8 weeks
  Mild depression (11-17 points) Moderate depression (18-29 points) Severe depression (30-63 points)
Visual Analogue Scale | 8 weeks
  To evaluate Fatigue. Each line is 100 mm in length - thus, scores fall between 0 and 100.Scoring : 0 : not all tired 100: extremely tired (left end of scale=not tired at all, right end of scale=extremely tired)
Quadriceps muscle strength | 8 weeks
  Muscle testing with dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided